CLINICAL TRIAL: NCT02752945
Title: Feasibility Randomised Controlled Trial of a One-day CBT Workshop ("DISCOVER") for 15-18 Year Olds With Anxiety and/or Depression in Clinic Settings
Brief Title: Feasibility Trial of a One-day CBT Workshop ("DISCOVER") for 15-18 Year Olds With Anxiety and/or Depression in Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 192806; 16/LO/0231 (Other: NHS Ethics Reference); R&D2016/021 (Other: NHS Trust approval)
Record Dates: First submitted 2016-04-14; First posted 2016-04-27 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2016-04

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Discover LC

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- One-day CBT workshop (+Usual Care) (Experimental): One-day CBT-based workshop ("DISCOVER"), followed by up to three brief telephone contacts to review goals set in workshop.
  Interventions: Other: One-day CBT workshop; Other: Usual care
- Usual care (Active Comparator): Usual care afforded by local CAMHS services
  Interventions: Other: Usual care

INTERVENTIONS:
Other: One-day CBT workshop — One-day long CBT workshop, with between 4-15 participants, facilitated by clinical psychologists. Following introductions, ice breakers and an explanation of the CBT model, CBT techniques are then introduced and practised using a variety of methods. One week after the workshop, any personal goals set during the workshop are reviewed with one of the workshop facilitators in a 'telephone goal review.'
  Other Names: DISCOVER
  Arms: One-day CBT workshop (+Usual Care)
Other: Usual care — Usual care afforded by local CAMHS services

SUMMARY:
This is a feasibility trial designed to test the feasibility and acceptability of a one-day Cognitive Behavioural Therapy (CBT) workshop intervention ("DISCOVER") for young people aged between 15-18 years, who are on local child and adolescent mental health services (CAMHS) waiting lists, awaiting treatment for difficulties with anxiety and/or depression. Participants will be randomised to receive either the DISCOVER workshop (in addition usual care) or to continue usual care.

DETAILED DESCRIPTION:
Sclare and colleagues (2015) have developed an open-access intervention ("DISCOVER") for 16-18 year olds experiencing emotional problems, in the form of one-day CBT-based workshops, delivered in schools. DISCOVER has been tested in schools and preliminary outcomes have shown to be positive. Given the lengthy waiting lists of some CAMHS services, the present study seeks to explore whether the DISCOVER programme can be implemented in clinic settings, with a broader age range of 15-18 year olds, with the aim of providing young people with some form of help, whilst they are awaiting more individualised treatment. Fifteen to eighteen year olds awaiting treatment for anxiety and/or depression will be recruited from local CAMHS waiting lists, and randomised to receive either the DISCOVER workshop, delivered in clinic (in addition to usual care), or to continue usual care. The study will assess the feasibility, acceptability and range of outcomes of DISCOVER in clinic settings.

ELIGIBILITY:
Inclusion Criteria:

1. aged 15-18 years;
2. fluent in English;
3. currently on a local CAMHS waiting list for treatment based on a referral for emotional difficulties (anxiety and/or depression);
4. willing and able to attend a one-day workshop within clinic; and
5. their position on the waiting list must indicate that they are unlikely to receive a CAMHS treatment appointment in the 8 weeks following the workshop.

Exclusion Criteria:

1. presenting with acute risk of harm to self or others;
2. have severe learning difficulties; and
3. are unable to provide informed written consent to participate and are unable to complete assessments.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mood and Feelings Questionnaire (MFQ) | 8 weeks
  Assesses symptoms of depression

SECONDARY OUTCOMES:
Revised Child Anxiety and Depression Scale (RCADS) | 8 weeks
  Assesses symptoms of anxiety
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | 8 weeks
  Assesses psychological well-being

CONTACTS AND LOCATIONS:
Overall Officials: Christina E Loucas, BSc, Principal Investigator — Institute of Psychiatry, Psychology & Neuroscience, King's College London
Locations (1):
- South London and Maudsley NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Loucas CE, Sclare I, Stahl D, Michelson D. Feasibility randomized controlled trial of a one-day CBT workshop ('DISCOVER') for 15- to 18-year-olds with anxiety and/or depression in clinic settings. Behav Cogn Psychother. 2020 Mar;48(2):142-159. doi: 10.1017/S1352465819000286. Epub 2019 May 20. PMID 31106728
- See also: Pubmed link — https://www.ncbi.nlm.nih.gov/pubmed/31106728
- See also: Study link — https://www.cambridge.org/core/journals/behavioural-and-cognitive-psychotherapy/article/feasibility-randomized-controlled-trial-of-a-oneday-cbt-workshop-discover-for-15-to-18yearolds-with-anxiety-andor-depression-in-clinic-settings/3ACAD61B1EFD4EC9750061828F312891